CLINICAL TRIAL: NCT06181812
Title: Prevalence of Pathogenic or Likely Pathogenic Germline Variants in Cancer Predisposition Genes Among Patients With Lung Adenocarcinoma
Brief Title: Pathogenic Variants in Genes Associated With Lung Adenocarcinoma
Status: Recruiting | Type: Observational
Sponsor: Oscar Gerardo Arrieta Rodríguez (Other)
Responsible Party: Sponsor-Investigator, Oscar Gerardo Arrieta Rodríguez, Coordinator of the Thoracic Oncology Unit and Laboratory of Personalized Medicine, Instituto Nacional de Cancerologia de Mexico
Organization: Instituto Nacional de Cancerologia de Mexico (Other)
Other Study IDs: (022/056/ICI)(CEI/057/22)
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Lung Adenocarcinoma
Keywords: Lung adenocarcinoma; Hereditary Cancer; Germline Pathogenic/Likely pathogenic variants; Somatic driver alterations
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — peripheral blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to describe the prevalence of germ line-pathogenic variants in Mexican patients with lung adenocarcinoma.

The main questions it aims to answer are:

1. What is the prevalence of pathogenic variants in genes associated with lung adenocarcinoma in Mexican patients younger than fifty?
2. Which clinical-pathological characteristics are associated with germ-line pathogenic variants in patients with lung adenocarcinoma?
3. How actionable somatic mutations are associated with germ line-pathogenic variants of patients with lung adenocarcinoma?

Participants will be asked to sign an informed consent; after that, they will be instructed to donate 10 ml of peripheral blood by venipuncture in the morning and before the patient has taken morning medication and the first meal, following a period of 8-12 hr fasting.

DETAILED DESCRIPTION:
This is an observational, descriptive, and longitudinal study.

The sample size was calculated with a proportion difference formula for a known population, considering the Local Institutional Personalized Medicine Laboratory tests 100 blood samples per year from patients with non-small cell lung cancer (NSCLC). It was considered a 95% confidence level and an 80% power. In addition, a 10% loss in follow-up was estimated.

After reviewing the inclusion and exclusion criteria, signing the informed consent, and peripheral blood sampling. Total DNA (tDNA) will be extracted using the DNAeasy Blood & Tissue (Qiagen) kit.

Likewise, for the determination of pathogenic variants, the Sophia HCS Community panels (Sophia genetics) will be used to carry out Next-generation (NGS) sequencing in a NextSeq 550 (Illumina) platform.

To determine the clinical significance of genomic variants, the data analysis will be performed on the SOPHiA Alamut™ Visual Plus which is a comprehensive, full genome browser for efficient and user-friendly variant interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* ≥ 16 years old, according the institutional protocols for new patients admittances.
* histologically confirmed lung adenocarcinoma (LUAD)
* Signed written informed consent form
* A life expectancy greater than 8 weeks.
* Histologically confirmed LUAD and one of the following conditions: i) LCFH, defined as having one first-degree relative (FDR) or two or more second-degree relatives with LC, irrespective of the age at diagnosis. ii) Age at diagnosis ≤50 years, or ≤60 with a pack-years index. iii) Presence of ≥1 AGAs (EGFR, ALK, ROS1, KRAS, BRAF, MET exon 14 skipping, or RET).

Exclusion Criteria:

* A sample of peripheral blood that is not accessible.
* Insufficient clinical pathological information in the electronic clinical record.

Elimination Criteria:

* Withdrawal
* Insufficient DNA quality and quantity for genomic sequencing analyses.
* Lost of follow up

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with lung adenocarcinoma treated in the Thoracic Oncology Unit of the National Institute of Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
PV in patients with lung carcinoma | One peripherial blood sample (day 1) at baseline of study.
  To determine the prevalence of pathogenic variants (PV) in patients with lung adenocarcinoma through amplicon next-generation sequencing (NGS).

SECONDARY OUTCOMES:
OS | From date of confirmed diagnosis until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To evaluate the prognostic impact of the pathogenic variants (PV) in the overall survival (OS) of patients with lung carcinoma.
PFS | From date of first line of treatment initiation (guided therapy) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  To evaluate the prognostic impact of the pathogenic variants (PV) in the progression free survival (PFS) of patients with lung carcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G Arrieta Rodriguez, M.D., M.Sc., Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- Thoracic Oncology Unit and Personalized Medicine Laboratory, Instituto Nacional de Cancerología, Mexico City, Mexico

REFERENCES:
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204
- [Background] Kumar R, Castillero F, Bhandari S, Malapati S, Kloecker G. The Hispanic Paradox in Non-Small Cell Lung Cancer. Hematol Oncol Stem Cell Ther. 2022 Jun 1;15(2):21-29. doi: 10.1016/j.hemonc.2021.02.004. PMID 33775613
- [Background] Mukherjee S, Bandlamudi C, Hellmann MD, Kemel Y, Drill E, Rizvi H, Tkachuk K, Khurram A, Walsh MF, Zauderer MG, Mandelker D, Topka S, Zehir A, Srinivasan P, Esai Selvan M, Carlo MI, Cadoo KA, Latham A, Hamilton JG, Liu YL, Lipkin SM, Belhadj S, Bond GL, Gumus ZH, Klein RJ, Ladanyi M, Solit DB, Robson ME, Jones DR, Kris MG, Vijai J, Stadler ZK, Amos CI, Taylor BS, Berger MF, Rudin CM, Offit K. Germline Pathogenic Variants Impact Clinicopathology of Advanced Lung Cancer. Cancer Epidemiol Biomarkers Prev. 2022 Jul 1;31(7):1450-1459. doi: 10.1158/1055-9965.EPI-21-1287. PMID 35477182
- [Background] Sorscher S, LoPiccolo J, Heald B, Chen E, Bristow SL, Michalski ST, Nielsen SM, Lacoste A, Keyder E, Lee H, Nussbaum RL, Martins R, Esplin ED. Rate of Pathogenic Germline Variants in Patients With Lung Cancer. JCO Precis Oncol. 2023 Sep;7:e2300190. doi: 10.1200/PO.23.00190. PMID 37992258
- [Background] Peng W, Li B, Li J, Chang L, Bai J, Yi Y, Chen R, Zhang Y, Chen C, Pu X, Jiang M, Li J, Zhong R, Xu F, Chen B, Xu L, Wang N, Huan J, Dai P, Guan Y, Yang L, Xia X, Yi X, Wang J, Yu F, Wu L. Clinical and genomic features of Chinese lung cancer patients with germline mutations. Nat Commun. 2022 Mar 10;13(1):1268. doi: 10.1038/s41467-022-28840-5. PMID 35273153
- [Background] Carrot-Zhang J, Soca-Chafre G, Patterson N, Thorner AR, Nag A, Watson J, Genovese G, Rodriguez J, Gelbard MK, Corrales-Rodriguez L, Mitsuishi Y, Ha G, Campbell JD, Oxnard GR, Arrieta O, Cardona AF, Gusev A, Meyerson M. Genetic Ancestry Contributes to Somatic Mutations in Lung Cancers from Admixed Latin American Populations. Cancer Discov. 2021 Mar;11(3):591-598. doi: 10.1158/2159-8290.CD-20-1165. Epub 2020 Dec 2. PMID 33268447
- [Background] Gerson R, Zatarain-Barron ZL, Blanco C, Arrieta O. Access to lung cancer therapy in the Mexican population: opportunities for reducing inequity within the health system. Salud Publica Mex. 2019 May-Jun;61(3):352-358. doi: 10.21149/10118. PMID 31276352
- [Background] Wang Y, McKay JD, Rafnar T, Wang Z, Timofeeva MN, Broderick P, Zong X, Laplana M, Wei Y, Han Y, Lloyd A, Delahaye-Sourdeix M, Chubb D, Gaborieau V, Wheeler W, Chatterjee N, Thorleifsson G, Sulem P, Liu G, Kaaks R, Henrion M, Kinnersley B, Vallee M, LeCalvez-Kelm F, Stevens VL, Gapstur SM, Chen WV, Zaridze D, Szeszenia-Dabrowska N, Lissowska J, Rudnai P, Fabianova E, Mates D, Bencko V, Foretova L, Janout V, Krokan HE, Gabrielsen ME, Skorpen F, Vatten L, Njolstad I, Chen C, Goodman G, Benhamou S, Vooder T, Valk K, Nelis M, Metspalu A, Lener M, Lubinski J, Johansson M, Vineis P, Agudo A, Clavel-Chapelon F, Bueno-de-Mesquita HB, Trichopoulos D, Khaw KT, Johansson M, Weiderpass E, Tjonneland A, Riboli E, Lathrop M, Scelo G, Albanes D, Caporaso NE, Ye Y, Gu J, Wu X, Spitz MR, Dienemann H, Rosenberger A, Su L, Matakidou A, Eisen T, Stefansson K, Risch A, Chanock SJ, Christiani DC, Hung RJ, Brennan P, Landi MT, Houlston RS, Amos CI. Rare variants of large effect in BRCA2 and CHEK2 affect risk of lung cancer. Nat Genet. 2014 Jul;46(7):736-41. doi: 10.1038/ng.3002. Epub 2014 Jun 1. PMID 24880342
- [Background] Esai Selvan M, Zauderer MG, Rudin CM, Jones S, Mukherjee S, Offit K, Onel K, Rennert G, Velculescu VE, Lipkin SM, Klein RJ, Gumus ZH. Inherited Rare, Deleterious Variants in ATM Increase Lung Adenocarcinoma Risk. J Thorac Oncol. 2020 Dec;15(12):1871-1879. doi: 10.1016/j.jtho.2020.08.017. Epub 2020 Aug 28. PMID 32866655